CLINICAL TRIAL: NCT04946006
Title: Maintenance Infusion of Oxytocin Following Elective Cesarean Deliveries: an Up-down Sequential Allocation Dose-response Study
Brief Title: Maintenance Infusion of Oxytocin Following Elective Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-05
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Hemorrhage
Keywords: Cesarean delivery; oxytocin; uterotonic; pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Biased coin up-and-down design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Oxytocin infusion rate 2 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 2 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 4 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 4 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 6 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 6 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 8 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 8 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 10 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 10 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 12 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 12 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 14 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 14 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 16 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 16 IU/h.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin will be prepared in a 1L bag of Ringer's lactate, to be infused at a rate of 125 ml/h.
  Other Names: Pitocin

SUMMARY:
This study is designed to determine the minimal effective oxytocin maintenance dose required during cesarean delivery to achieve the best effect. Oxytocin is a drug which is routinely used to help contract the uterus and keep it contracted after the delivery of the baby and placenta. The aim of oxytocin is to reduce the amount of blood that might be lost. In order to determine the minimal effective dose, the investigators will conduct a dose-finding study. The first patient will receive a set oxytocin infusion. If the uterus contracts well, this is considered satisfactory and the next patient will receive the same dose. If the uterus does not contract well, this is considered unsatisfactory and the next patient will receive a higher dose. The dose for the next patient will be determined based on the results of the uterine contraction of the previous patient.

The investigators hypothesize that the ED90 of an oxytocin infusion rate to maintain a satisfactory uterine tone during a cesarean delivery in non-laboring women, would be lower than that found in previous studies without an initial bolus (less than 16 IU/h).

DETAILED DESCRIPTION:
This study will be conducted as a prospective, double blinded clinical trial (patient, anesthesiologist and obstetrician blinded to the oxytocin dose), in an up-down sequential allocation fashion. The objective of the study is to determine the minimum effective dose of oxytocin infusion required to produce appropriate uterine contraction during and after cesarean delivery under neuraxial anesthesia in non-laboring women. For the purpose of this study, the minimum effective dose is defined to be that at which adequate response occurs in 90% of patients, i.e. ED90.

ELIGIBILITY:
Inclusion Criteria:

* Elective uncomplicated cesarean delivery under neuraxial anesthesia
* >18 year-old with ASA status II or III, with a singleton gestation and a gestational age between 37 to 42 weeks Informed consent to participate in this study

Exclusion Criteria:

* Refusal to give written informed consent
* Allergy or hypersensitivity to oxytocin
* Body mass index ≥ 40 kg/m2on the day of admission
* A history of hypertension and/ or severe cardiac disease(s)
* Contra-indications for neuraxial anesthesia
* Conditions that predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, preeclampsia, macrosomia (≥ 4 kg), polyhydramnios, uterine fibroids in and near operating field, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Uterine tone upon discharge from the post anesthetic care unit (PACU): questionnaire | 2 hours
  Uterine tone will be evaluated as satisfactory or unsatisfactory by the obstetrician throughout the surgery, starting at 5 minutes after the oxytocin infusion. It will also be measured at 10 minutes following the oxytocin infusion and every 10 minutes following that for the duration of the surgery. Unsatisfactory uterine tone at any time until discharge from the PACU will be considered a failure of the maintenance infusion.

SECONDARY OUTCOMES:
Calculated blood loss | 24 hours
  Estimated blood loss will be calculated using the difference in hematocrit values prior to surgery and 24 hours post surgery, using the following formula:
  Calculated blood loss (mL) = EBV ((Pre-op Htc-Post-op Htc)/pre-op Htc) EBV (estimated blood volume) in ml: patient's weight in kg x 85.
Incidence of post partum hemorrhage | 24 hours
  Incidence of post partum hemorrhage defined as a calculated blood loss >1L.
Need for blood transfusion | 24 hours
  Blood product administered.
Episodes of bleeding postpartum | 24 hours
  Number of episodes of bleeding postpartum up to 24 hours post delivery.
Intraoperative requirement for additional uterotonic medication | 2 hours
  A request made by the obstetrician performing the cesarean delivery for additional uterotonic medication, due to bleeding or poor uterine tone.
Requirement for additional uterotonic medication in the PACU | 2 hours
  Any uterotonic medication administered while the patient is in PACU
Requirement for additional uterotonic medication from discharge from the PACU until 24 hours postpartum. | 24 hours
  Any uterotonic medication administered after the patient is discharged from PACU until 24 hours postpartum.
Postoperative uterine position in the PACU | 3 hours
  Postoperative uterine position (below or above the umbilicus) as determined by the PACU nurse. This is measured every 15 minutes for the first hour and then hourly until discharge to the postpartum unit.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Hypertension: systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline or a heart rate < 50bpm, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Boonstra L, Carvalho JCA, Turner W, Downey K, Ye XY, Thomas J, Balki M. Maintenance infusion rate of oxytocin after initial 1-IU bolus for elective Cesarean delivery: a dose-finding study. Can J Anaesth. 2024 Oct;71(10):1363-1371. doi: 10.1007/s12630-024-02828-9. Epub 2024 Sep 19. PMID 39300008